CLINICAL TRIAL: NCT05910528
Title: A Phase 2, Multicenter, Double-blind, Two-arm Study of Subcutaneous RO7790121 for the Treatment of Subjects With Moderate to Severe Active Crohn's Disease
Brief Title: Afimkibart (RO7790121) for the Treatment of Moderate to Severe Active Crohn's Disease
Acronym: TAHOE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA45392; 2023-504265-23-00 (EU CTIS Number); NCT06370858 (obsolete NCT alias)
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Crohns Disease
Keywords: Crohns Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence A; Drug: Afimkibart (RO7790121) Induction dose A, Maintenance dose and OLE dose (Experimental)
  Interventions: Drug: Afimkibart
- Treatment Sequence B; Drug: Afimkibart (RO7790121) Induction dose B, Maintenance dose and OLE dose (Experimental)
  Interventions: Drug: Afimkibart

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered during the Induction, Maintenance and OLE period.
  Other Names: RO7790121; RVT-3101; PF-06480605

SUMMARY:
This Phase 2, randomized, double-blind, multicenter, induction and maintenance study is designed to evaluate the safety and efficacy of Afimkibart (RO7790121, RVT-3101) in adult participants with moderate to severe active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Moderately to severely active CD as defined by CDAI and SES-CD, assessed by central read
* Elevated very soft or liquid stool frequency and/or abdominal pain
* Must have no response, insufficient response, loss of response and/or intolerance to at least 1 conventional therapy (e.g. corticosteroids) or advanced therapy

Exclusion Criteria:

* Diagnosis of ulcerative colitis, indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis or active diverticular disease
* Short gut syndrome
* Presence of an ostomy or ileoanal pouch
* Bowel resection or diversion with ~6-months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAE), Serious Adverse Events (SAE) and AE Leading to Discontinuation | Until end of study, approximately 5 years

SECONDARY OUTCOMES:
Proportion of Participants Achieving Endoscopic Response | Week 14
  Endoscopic response defined as decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) >=50% from Baseline at Week 14
Proportion of Participants Achieving Clinical Remission by Crohn's Disease Activity Index (CDAI) | Week 14
  Clinical remission defined as CDAI <150 at Week 14
Proportion of Participants Achieving Clinical Remission by Patient Reported Outcome 2 (PRO2) | Week 14
  Clinical remission by PRO2 defined as average daily very soft or liquid stool frequency (SF) <= 2.8 and abdominal pain (AP) score <=1, and not worse than Baseline at Week 14.
Trough Concentration (Ctrough) | Up to Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (5):
  - Digestive Health Specialists, Dothan, Alabama
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - I.H.S Health Northwell Health, Kissimmee, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
- AZ Delta, Roeselare, Belgium
- France (3):
  - CHU de Nantes, Nantes
  - Institut des MICI, Clinique Ambroise Paré, Neuilly-sur-Seine
  - CHRU de Nancy Brabois, Vandœuvre-lès-Nancy
- Poland (2):
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing